CLINICAL TRIAL: NCT01437748
Title: Small Airways Evaluation and Peripherical Effect of Two Bronchodilators in Healthy Subjects and Stable COPD Patients
Brief Title: Closing Volume Interpretation and Bronchodilators Effect
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Milan (Other)
Collaborators: Fondazione Salvatore Maugeri (Other)
Responsible Party: Principal Investigator, Pierachille Santus, Head of Respiratory Rehabilitation Unit, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 629CEC
Record Dates: First submitted 2011-09-12; First posted 2011-09-21 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Healthy; COPD
Keywords: Small Airways; Closing volume; Closing Capacity; Tiotropium; Indacaterol; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Indacaterol maleate (Experimental): Indacaterol 300 mcg via Breezehaler Inhaler will be administered by a third independent investigator not involved in the performing of any of the tests decribed, following a randomization list
  Interventions: Drug: Indacaterol maleate
- Tiotropium bromide (Active Comparator): Tiotropium 18 mcg, via HandiHaler inhaler will be administered by a third independent investigator not involved in the performing of any of the tests decribed, following a randomization list
  Interventions: Drug: Tiotropium bromide

INTERVENTIONS:
Drug: Indacaterol maleate — Dry powder, 300 mcg, only one inhalation with 24 hours duration
  Other Names: Onbrez, Hirobriz, Onbrize, Oslif Breezehaler, Arcapta
  Arms: Indacaterol maleate
Drug: Tiotropium bromide — Dry powder, 18 mcg, only one inhalation with 24 hours duration
  Other Names: Spiriva
  Arms: Tiotropium bromide

SUMMARY:
* The gold standard measures to evaluate small airways (SAW) "in vivo" is not well understood
* Two tests are today used to measure SAW but real results concordance is not clear
* These problems have a small evidence
* Data about real effect of bronchodilators on SAW (eg Tiotropium and Indacaterol) has never been studied
* Only an acute bronchodilators effect, after one hour of drugs inhalation, will be evaluated
* The time frame of study evaluations per patient will be of three hours: one hour for basal test; one hour rest after drug administration; one hour for post bronchodilators test
* All enrolled subjects will be outpatients and will be evaluated after 24 hours of inhalatory drugs washout

DETAILED DESCRIPTION:
Evaluation of small airways both in healthy and Chronic Obstructive Pulmonary Disease (COPD)subjects still today remains a big problem with implications in diagnostic and clinical management. The first lung alteration in smokers is the bronchiolitis and possibility to understand real damage on this anatomical district should be very interesting. The first point of the study will be the SAW evaluation. The two principal technics to do this are: Single Breath Test (SBT) and oesophageal balloon (EB). With SBT is possible to obtain the four expiration phases and so the shift from phase 3 to phase 4 identifying the point called closing capacity (CC). With EB is possible to obtain the lung static pressure-volume curve and after this to identify the point of closing volume (CV). The real concordance of CC and CV has never been studied both in healthy and COPD subjects.

The SBT is performed by pneumotachograph matched with a gas analyzer. Patient breath normally for some seconds, exhales to residual volume (RV) and after that deeply inhales oxygen (100%) to total lung capacity (TLC), then the patient exhales slowly to RV. This test will be repeated a minimum of three times.

The evaluation of CV will be performed by EB. The oesophageal balloon is introduced by nose and located in distal oesophageal tract. By pressure transducer the correct position will be confirmed. After the investigators will perform the evaluation of lung volume, trans pleural pressure and flow. These parameters will be registered at tidal volume, during forced expiration and finally during hyperventilation.

So, after the identification of presence,absence and eventually concordance of CC and CV should be interesting to evaluate the possible effect on SAW of bronchodilators usually used in clinical practice. More in detail, the investigators will administered in random order and after basal evaluation of CV and CC dry powder of indacaterol 300 micrograms (mcg) or Tiotropium 18 mcg. After one hour of drug administration the investigators will repeat the maneuver for CC and CV evaluations. In this way, will be evaluated only the acute effect of the bronchodilators on lung hyperinflation. Each subjects will perform plethysmographic test too. Bronchodilators will be administered only to the COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Signature of informed consent
* Healthy subjects with age from 20 to 80 yars old and never smokers
* COPD diagnosis
* COPD with age from 50 to 85 years old
* History of COPD at least of noe year
* Respiratory stable conditions at least of one month
* Any basal FEV1 expressed in % of predicted value
* FEV1/Forced Vital Capacity (FVC) less than 70%
* COPD with history of former or active smokers with minimum of 20 pack year

Exclusion Criteria:

* Pregnancy
* FEV1/FVC more than 70%
* Known deficit of alpha 1 antitrypsin
* Subjects submitted to a Lung Volume Reduction Surgery (LVRS)
* Subjects with known positivity to Human Immunodeficiency Virus (HIV)
* Known intolerance to a nasogastric balloon
* Misuse of alcool or drugs
* Absence of compliance in performing respiratory test

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Closing Volume (CV) | Participants will be followed for the duration of medical office stay an expected average of 3 hours. The outcome measure will be assessed for the end of october 2011 and will be presented within december 2011.
  The evaluation of CV will be performed by EB. The oesophageal balloon is introduced by nose and located in distal oesophageal tract. By pressure transducer the correct position will be confirmed. After the investigators will perform the evaluation of lung volume, trans pleural pressure and flow. These parameters will be registered at tidal volume, during forced expiration and finally during hyperventilation.
Closing Capacity (CC) | Participants will be followed for the duration of medical office stay an expected average of 3 hours. The outcome measure will be assessed for the end of october 2011 and will be presented within december 2011
  The evaluation of CC will be measuired by Single Breath Test (SBT) and performed by pneumotachograph matched with a gas analyzer. Patient breath normally for some seconds, exhales to residual volume (RV) and after that deeply inhales oxygen (100%) to total lung capacity (TLC), then the patient exhales slowly to RV. This test will be repeated a minimum of three times.

SECONDARY OUTCOMES:
Effect of Tiotropium or Indacaterol on CV and CC registration | Participants will be followed for the duration of medical office stay an expected average of 3 hours. The outcome measure will be assessed for the end of october 2011 and will be presented within december 2011
  Possible effect on small airways by two distinct ultra long acting bronchodilators
Comparison concordance of CV and CC | Participants will be followed for the duration of medical office stay an expected average of 3 hours. The outcome measure will be assessed for the end of october 2011 and will be presented within december 2011
  This data will be important to identify the best, easiest and most reliable test for clinical SAW evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Pierachille Santus, MD, PhD, Study Director — Università degli Studi di Milano-Pneumologia Riabilitativa-Fondazione Salvatore Maugeri-MILANO
Locations (1):
- Pneumologia Riabilitativa-Fondazione Maugeri-Istituto Scientifico di Milano- IRCCS, Milan, Milano, Italy